CLINICAL TRIAL: NCT06308640
Title: Evaluation of Maxillary Molar Distalization With Two Bone Supported Protocols Using Cone Beam Computed Tomography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nouran Mohamed Abdelwahab Eissa, Assisstant Lecturer,Orthodontic Department,Faculty of Dentistry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORTH 11-23 2097
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Class II Malocclusion
Keywords: Molar Distalization; Fast Back Distalizer; Leaf Spring Self-Activated Expander
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to evaluate and compare the treatment effects of two bone supported protocols for bilateral distalization of maxillary molars in patients exhibiting class II pattern using Fast Back appliance and modified Leaf Spring Self-Activated Expander
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast Back Rapid Distalizer (Experimental): Group 1: Consisted of 10 patients, their upper molar will be distalized with bone suppored Fast Back (Fast Back Rapid Distalizer, leone, s.p.a, Italy).
  Interventions: Device: Insertion of the device intraorally
- Modified Leaf Spring Self-Activated Expander (Experimental): Group 2: Consisted of 10 patients, their upper molar will be distalized with bone supported modified Leaf Spring Self-Activated Expander. (Leaf Self Expander, leone, s.p.a, Italy).
  Interventions: Device: Insertion of the device intraorally

INTERVENTIONS:
Device: Insertion of the device intraorally — * The distalizer appliance will be checked for adaptation intraorally, the two bands of the maxillary first molars will be fitted in their accurate position on the teeth.
  * The screw insertion will be carried out with the patient under local anesthesia.
  * They will be placed inside the two eyelets of the anterior arms of the screw in the appliance

SUMMARY:
The goal of this clinical trial is to to evaluate and compare the skeletal and dental changes of bone supported Fast Back and bone supported modified Leaf Spring Self-Activated Expander in bilateral distalization of maxillary molars using CBCT in Egyptian people. The main question it aims to answer are: • If bone supported Fast Back and bone supported modified Leaf Spring Self-Activated Expander will be effective in bilateral distalization of maxillary molars

The patients will be selected according to the following criteria:

1. Patient with full permanent dentition.
2. Good oral hygiene.
3. None of the patients had received any orthodontic treatment.
4. Class II molar relationship.
5. Minimal or no crowding in the mandibular arch.
6. Non-extraction treatment plan with molar distalization.
7. Low angle cases.
8. No medical problems or active periodontal disease.

Researchers will compare between bone supported Fast Back appliance and bone supported modified Leaf Spring Self-Activated and see if they will be effective in maxillary molars distalization.

DETAILED DESCRIPTION:
The patients will be divided into two groups:

Group 1: Consisted of 10 patients, their upper molar will be distalized with bone suppored Fast Back (Fast Back Rapid Distalizer, leone, s.p.a, Italy).

Group 2: Consisted of 10 patients, their upper molar will be distalized with bone supported modified Leaf Spring Self-Activated Expander. (Leaf Self Expander, leone, s.p.a, Italy).

* Assessment of the 3D dentoskeletal treatment effects of the palatally bone supported Fast Back and palatally bone supported modified Leaf Spring Self-Activated Expander will be performed by using the CBCT scans.
* Pretreatment CBCT (T1) and post-distalization until study completion with an average of 1 year (T2) for each subject

All data will be collected, tabulated and statistically analyzed using the SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Patient with full permanent dentition.
* Good oral hygiene.
* Class II molar relationship.
* Non-extraction treatment plan with molar distalization.
* Low angle cases.
* medical problems or active periodontal disease.

Exclusion Criteria:

* The patients had received any orthodontic treatment.
* Crowding in the mandibular arch.
* Medical problems or active periodontal disease.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
3D Dental and skeletal Cephalometric Measurements | Through study completion, an average of 1 year"
  Using CBCT 3D Analysis
2D Dental and skeletal Cephalometric Measurements | Through study completion, an average of 1 year"
  Using CBCT 2D Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Safaa M Gaballah, Professor, Principal Investigator — Tanta University; Shaimaa M Elmarhoumy, professor, Study Director — Tanta University
Locations (1):
- Faculty of Dentistry, Tanta, Gharbia Governorate, Egypt